CLINICAL TRIAL: NCT04691128
Title: Comparison of Desflurane and Propofol for Brain Relaxation in Patients Undergoing Supratentorial Craniotomy：a Randomized Controlled Study
Brief Title: Desflurane and Brain Relaxation in Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H199510180629
Record Dates: First submitted 2020-12-12; First posted 2020-12-31 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Supratentorial Tumor
MeSH Terms: conditions — Supratentorial Neoplasms | interventions — Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane inhalational anesthesia (Experimental)
  Interventions: Drug: Desflurane
- Propofol total intravenous anesthesia (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Desflurane — After induction, anesthesia will be maintained with 0.8-1.3 MAC desflurane and 0.05-0.2 μg/kg/min remifentanil.
  Other Names: inhalational anesthesia
  Arms: Desflurane inhalational anesthesia
Drug: Propofol — After induction, anesthesia will be maintained with 6-8 mg/kg/h propofol and 0.05- 0.2 μg/kg/min remifentanil
  Other Names: TIVA; total intravenous anesthesia
  Arms: Propofol total intravenous anesthesia

SUMMARY:
Optional brain relaxation improves the surgeon's operating conditions and is likely to minimize the degree of retraction injury ,with the potential for providing patients with a better outcome. The choice of anesthetic drugs can affect intraoperative brain relaxation. Propofol suppresses brain metabolism, reduces cerebral blood flow, and provides satisfactory brain relaxation. Desflurane is often criticized in neurosurgery due to its cerebral vasodilation and potential to increase intracranial pressure, however, it has been found to have a little clinical significance. This study intends to compare the effects of desflurane with propofol on brain relaxation in patients with supratentorial tumors under mild hyperventilation, and to provide new clinical evidence for the use of desflurane in neurosurgical anesthesia.

DETAILED DESCRIPTION:
To compare the effect of desflurane versus propofol combined with remifentanil anesthesia on brain relaxation in patients undergoing supratentorial tumor surgery with mild hyperventilation, and compare the emergence time and common complications during recovery.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years
* Scheduled for elective craniotomy for supratentorial cerebral tumors
* ASA status I-III
* Glasgow score of 15
* No clinical signs of intracranial hypertension
* Preoperative brain imaging (CT or MRI) with midline shift less than 5mm
* Informed consent signed by patients

Exclusion Criteria:

* Scheduled intraoperative motor evoked potential monitoring
* Patients with cerebral vascular diseases
* Uncontrolled cardiopulmonary disease
* Schedule to retain tracheal intubation after surgery
* Unable to comprehend and cooperate with the examination
* BMI > 30 Kg/m-2
* Emergency surgery
* History of related anesthetic allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of satisfactory brain relaxation | during surgery
  Assessed by the neurosurgeon using a 4-point scale (1= perfectly relaxed, 2= satisfactorily relaxed, 3= firm brain, 4=bulging brain) at the opening of the dura mater, score 1 and 2 represent satisfactory brain relaxation

SECONDARY OUTCOMES:
Emergence time | from drug discontinuation to eye opening, assessed up to 1 hours
  from drug discontinuation to eye opening
Extubation time | from drug discontinuation to tracheal extubation, assessed up to 1 hours
  from drug discontinuation to tracheal extubation
Postoperative complications | from drug discontinuation to discharge from PACU (Postanesthesia care unit), assessed up to 3 hours
  incidence of hypoxemia, hypotension, hypertension, tachycardia, bradycardia, agitation, shivering.
Postoperative pain and postoperative nausea and vomiting (PONV) | during the PACU stay and postoperative day 1.
  evaluated by Visual Analogue Score(VAS).
Duration in PACU (Postanesthesia care unit) | from entering PACU to exiting PACU, an expected average of 1 hour
  time from entering PACU to exiting PACU
Early postanesthesia cognitive recovery | at 15, 30min after tracheal extubation
  evaluated by Short Orientation Memory Concentration Test (SOMCT)
Dural tension | during surgery
  evaluated using a 4-point scale after bone flap removal.
Quality of anesthesia recovery | at postoperative day 1
  assessed by quality of recovery-15 scale (QoR-15)
Anesthesia expenses | at postoperative day 1
  Total cost of anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Jiang Z, Wu Y, Liang F, Jian M, Liu H, Mei H, Han R. Brain relaxation using desflurane anesthesia and total intravenous anesthesia in patients undergoing craniotomy for supratentorial tumors: a randomized controlled study. BMC Anesthesiol. 2023 Jan 10;23(1):15. doi: 10.1186/s12871-023-01970-z. PMID 36624384